CLINICAL TRIAL: NCT06047197
Title: Phase I Clinical Trial of Dinorencel Injection (or RC19D2 Cell Injection) in the Treatment of CD19-positive Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: Phase I Clinical Trial of RC19D2 Cell Injection in the Treatment of Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Yongtai Ruike Biotechnology Company Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC19D2-r/r DLBCL-01
Record Dates: First submitted 2023-09-01; First posted 2023-09-21 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-cell Lymphoma
Keywords: CD19; CAR-T; RC19D2; DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First dose group (Experimental): The initial dose is (0.5 ± 0.1) × 10^6/kg, with 1 participant enrolled
  Interventions: Biological: RC19D2 cell injection
- Second dose group (Experimental): The second dose is (1.0 ± 0.2) × 10^6/kg, with 3-6 study participants enrolled
  Interventions: Biological: RC19D2 cell injection
- Third dose group (Experimental): The third dose is (2.5± 0.5) × 10^6/kg, with 3-6 study participants enrolled
  Interventions: Biological: RC19D2 cell injection
- Fourth dose group (Experimental): The fourth dose is (5± 1) × 10^6/kg, with 3-6 study participants enrolled
  Interventions: Biological: RC19D2 cell injection

INTERVENTIONS:
Biological: RC19D2 cell injection — The functional component of RC19D2 cell injection is T cells that have been genetically modified to express anti CD19 chimeric antigen receptors.

SUMMARY:
This trial is a phase I clinical trial aimed at the safety and tolerability of RC19D2 cell injection in the treatment of CD19 positive patients with recurrent or refractory diffuse large B-cell lymphoma

DETAILED DESCRIPTION:
This trial is a Phase I clinical trial, which is divided into two trial stages. The first stage is a dose-increasing trial stage The second stage is the dose extension experiment stage.

The main endpoint is to evaluate its tolerance and safety. The first dose group used rapid titration method for dose increase, and the subsequent dose groups used the classic 3+3 experimental design for dose increase. A total of 4 dose groups are planned to be set up. The second to fourth dose groups will include 3-6 participants in each group

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign the informed consent form;
* Age ≥ 18 years old at the time of screening, regardless of gender;
* Patients with diffuse large B-cell lymphoma who have been diagnosed as CD19 positive by histopathology and/or cytology, but have failed standard treatment in the early stage, and currently lack effective treatment methods for recurrent or refractory CD19 positive.
* The regulations for the past treatment status of research participants are as follows (meeting at least one of them): 1.At least after sufficient second-line treatment (CD20 positive individuals must have already used sufficient amounts of CD20 targeted drugs and anthracycline drugs), recurrence, no remission, or progression; In the first two lines of treatment, if the optimal therapeutic effect is SD, then the line of treatment must have completed 2 cycles;2.Recurrence, unrelieved, or progression after autologous hematopoietic stem cell transplantation;
* According to the 2023 NCCN Lymphoma Treatment Guidelines and the 4th edition of the WHO Lymphatic Tissue Tumor Classification in 2016, the following types were included in this trial:Diffuse large B-cell lymphoma (DLBCL) non-specific (DLBCL-NOS)；Transforming follicular lymphoma (tFL)；High grade B-cell lymphoma (HGBL) with MYC, BCL2, and/or BCL6 rearrangement；High grade B-cell lymphoma, non-specific (HGBL-NOS)；Primary mediastinal large B-cell lymphoma (PMBL)；Grade 3b follicular lymphoma (FL3b);
* Expected survival time ≥ 12 weeks;
* There are measurable target lesions in imaging: the length and diameter of lesions in lymph nodes ≥ 15mm, or extranodal lesions>10mm (according to Lugano2014 standard); Lesions that have received radiotherapy in the past are considered measurable only when there is clear progress after completing radiotherapy;
* During screening, laboratory inspections must meet the following requirements:Neutrophil count ≥ 1.0 × 10^9/L;Lymphocyte count ≥ 0.3 × 10^9/L; Hemoglobin ≥ 70 g/L;Platelets ≥ 50 × 10^9/L;Total serum bilirubin ≤ 2.0 × Upper limit of normal value (ULN);Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN;Creatinine<1.5 × ULN and endogenous creatinine clearance rate ≥ 60 mL/min (creatinine clearance rate Cockcroft Fault method: male creatinine clearance rate=[(140 age) × Weight (kg)]/[0.818 × Creatinine（ μ Mol/L)]; Female creatinine clearance rate=[(140 age) × Body weight (kg) × 0.85]/[0.818 × Creatinine（ μ Mol/L)].
* The lung function is good, and the blood oxygen saturation of the fingertip pulse under non oxygen inhalation is ≥ 92%;
* The Eastern Oncology Collaborative Group (ECOG) physical fitness score is 0 or 1;
* Head MRI shows no central nervous system lymphoma;
* Cardiac ultrasound shows left ventricular ejection fraction ≥ 50%; No clinically significant abnormal electrocardiogram findings; No clinically significant pericardial or pleural effusion;
* Adequate venous access (for single collection) and no other contraindications for blood cell separation;
* The screening period blood pregnancy test for female participants of childbearing age must be negative

Exclusion Criteria:

* Individuals with a history of allergies to any component in cellular products;
* Individuals with a history of allogeneic hematopoietic stem cell transplantation;
* Individuals with a history of organ transplantation;
* hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg) are positive; Hepatitis B e antibody (HBe Ab) and/or hepatitis B core antibody (HBc Ab) are positive, and the HBV-DNA quantity is higher than the upper limit of normal value; Hepatitis C virus antibody (HCV Ab) is positive and HCV RNA quantification is higher than the upper limit of normal values; Positive for human immunodeficiency virus antibody (HIV-Ab); Positive anti Treponema pallidum antibody (TP Ab); Cytomegalovirus DNA quantification is higher than the upper limit of normal values; EB virus DNA quantification is higher than the upper limit of normal values;
* CNS diseases that have clinical significance in the past or screening, such as epilepsy, epileptic seizures, paralysis, aphasia, cerebral vascular ischemia/bleeding, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, mental illness, etc;
* Patients with active primary or secondary central nervous system (CNS) lymphoma (patients with CNS disease symptoms must undergo lumbar puncture examination to rule out CNS lymphoma).
* Those who have previously received other genetically modified T cell therapies, or other CAR-T therapies, or any other targeted therapy against CD19;
* Having severe genetic or autoimmune diseases (such as systemic lupus erythematosus);
* Screening for thromboembolic events within the first 6 months (such as myocardial infarction, pulmonary infarction, deep vein thrombosis, and other systemic thrombotic diseases);
* Screening for malignant tumors other than those indicated in this study within the first 5 years, except for tumors in situ (such as cervical cancer, bladder, breast cancer) or non melanoma skin cancer;
* Active or uncontrollable infections that require systemic treatment;
* Within 9 months prior to PBMC collection, received treatment with Bendamustine、Alenzumab, Fludarabine,and Cladribine;;
* Within 4 weeks prior to PBMC collection, patients received naloxamine, calcineurin inhibitors, chemotherapy drugs (methotrexate, cyclophosphamide, ifosfamide, benzoate nitrogen mustard or mefalam,), mycophenolate, thalidomide, immunosuppressive antibodies such as anti TNF, anti IL6, or anti IL6R therapy, tumor radiotherapy, or drugs that can bind to FKBP 12 protein (such as rapamycin, tacrolimus, everolimus, etc.);
* Long acting cell growth factors (such as polyethylene glycol recombinant human granulocyte stimulating factor PEG-rhG-CSF) were used within 3 weeks prior to PBMC collection;
* Received granulocyte macrophage colony stimulating factor (GM-CSF) treatment within 2 weeks prior to PBMC collection;
* Individuals who have received short-term cell growth factors (such as recombinant human granulocyte colony-stimulating factor, recombinant human thrombopoietin, etc.), hematopoiesis agonists/stimulators (such as haitrapopa ethanolamine tablets), CD20 monoclonal antibodies, and corticosteroids within 7 days prior to PBMC collection (excluding those who have received inhaled, local steroid therapy, and physiological replacement therapy for adrenal insufficiency);
* Received platelet transfusion within 7 days before the screening period;
* Pregnant or lactating women, or men or women with fertility potential, refuse to use contraception during the trial period and at the end of the trial (2 years after RC19D2 cell reinfusion);
* Patients who have participated in other drug clinical trials within 4 weeks prior to PBMC collection (new drug clinical trials, registered studies, clinical studies initiated by researchers, etc.);
* The researcher believes that this clinical trial is not suitable (such as poor compliance, drug abuse, etc.);
* Those who have received live or attenuated vaccines within 3 months prior to PBMC collection, or are expected to need to receive such vaccines during this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-09-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
MTD | 28 days
  Determine the maximum tolerable dose(MTD) based on the 28 day dose limit toxicity occurrence of all participants.
AE Safety | 2 years
  Number of participants with Adverse event (AESI, ADR, SAE, etc.), with abnormal laboratory test results, abnormal vital signs, abnormal physical examination findings and abnormal 12 lead electrocardiogram readings

CONTACTS AND LOCATIONS:
Overall Officials: lugui Qiu, MD, Principal Investigator — blood diseases hospital，chinese academy of medical sciences
Locations (1):
- Hematology Hospital of the Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China